CLINICAL TRIAL: NCT07308860
Title: Fractional Flow Reserve Versus Angiography for Multivessel Evaluation (FAME) 3 Extended A Comparison of Fractional Flow Reserve-Guided Percutaneous Coronary Intervention and Coronary Artery Bypass Graft Surgery in Patients With Multivessel Coronary Artery Disease
Brief Title: Fractional Flow Reserve Versus Angiography for Multivessel Evaluation (FAME) 3 Extended
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, William Fearon, MD, Professor of Medicine, Stanford University
Other Study IDs: 83374; 1R01HL179196-01 (NIH)
Record Dates: First submitted 2025-12-19; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
Keywords: CABG; FFR-guided PCI; quality of life; repeat revascularization; long term mortality; 3-vessel CAD; angina; 10-year mortality; stroke; cardiac death; stent; PCI; myocardial infarction; multicenter; coronary artery bypass; clinical trial; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Stroke; Death; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FFR-guided PCI group: These patients have undergone fractional flow reserve-guided percutaneous coronary intervention
  Interventions: Procedure: FFR-guided PCI
- CABG group: These patients underwent coronary artery bypass grafting surgery
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: FFR-guided PCI — Coronary stenting compared with coronary bypass surgery
  Groups: FFR-guided PCI group
Procedure: CABG — Coronary artery bypass surgery
  Groups: CABG group

SUMMARY:
Coronary artery disease, or narrowing of the blood vessels that provide blood to the heart, is the most common cause of death in the United States and can be treated with either coronary bypass surgery or coronary stent placement. This study will evaluate outcomes, including death and quality of life, at 10 years in 1,500 patients with coronary disease who have already been randomized to either bypass surgery or stenting.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains the major cause of morbidity and mortality in adults in the United States. In patients with 3-vessel CAD not involving the left main coronary artery, percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG) can improve outcomes. Older studies have shown that the more invasive option, CABG, significantly reduces mortality during long-term follow-up compared with PCI. However, these studies did not use contemporary methods to perform PCI, such as measuring an index called fractional flow reserve (FFR) with a coronary pressure wire or using current- generation drug-eluting stents (DES), both of which significantly improve outcomes after PCI. The Fractional flow reserve versus Angiography for Multivessel Evaluation (FAME) 3 trial randomized 1,500 patients to FFR-guided PCI with current generation DES or to CABG and found that at 5 years there was no significant difference in the composite of death, myocardial infarction (MI) or stroke between the two strategies. There was a reduction in MI in the CABG group. Longer-term follow-up is critical to determine if contemporary PCI results in similar survival as CABG. The primary aim of this project is to determine if 10-year mortality is different after FFR-guided PCI compared with CABG. Investigators will perform 10-year follow-up in the 1,500 patients randomized in the FAME 3 trial to determine if FFR-guided PCI is non-inferior to CABG with respect to mortality. Secondary aims include assessing quality of life and angina relief at 10 years in the two groups. Additionally, investigators will compare individual rates of secondary clinical outcomes including MI, stroke, and repeat revascularization at 10-year follow-up after PCI or CABG.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years with angina and/or evidence of myocardial ischemia
2. Three vessel CAD, defined as ≥ 50% diameter stenosis by visual estimation in each of the three major epicardial vessels or major side branches, but not involving left main coronary artery, and amenable to revascularization by both PCI and CABG as determined by the Heart Team. Patients with a non-dominant right coronary artery may be included if only the left anterior descending artery (LAD) and left circumflex have

   ≥50% stenosis
3. Willing and able to provide informed, written consent

Exclusion Criteria:

1. Requirement for other cardiac or non-cardiac surgical procedure (e.g., valve replacement, carotid revascularization), however a maze procedure or pulmonary vein isolation is allowed
2. Cardiogenic shock and/or need for mechanical/pharmacologic hemodynamic support
3. Recent STEMI (<5 days prior to randomization)
4. Ongoing Non STEMI with biomarkers (cardiac troponin) still rising
5. Known left ventricular ejection fraction <30%
6. Life expectancy < 2 years
7. Requiring renal replacement therapy
8. Undergoing evaluation for organ transplantation
9. Participation or planned participation in another clinical trial, except for observational registries
10. Pregnancy
11. Inability to take dual antiplatelet therapy or anticoagulation and single antiplatelet therapy for at least six months
12. Previous CABG
13. Left main disease requiring revascularization
14. Extremely calcified or tortuous vessels precluding FFR measurement
15. Any target lesion with in-stent drug-eluting stent restenosis
16. More than one major epicardial vessel which is chronically occluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will evaluate outcomes, including death and quality of life, at 10 years in 1,500 patients with coronary disease who have already been randomized to either bypass surgery or stenting.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival | 10-year follow-up
  The primary outcome is mortality or overall survival

SECONDARY OUTCOMES:
Quality of life | 10-year follow-up
  Secondary aims include assessing quality of life at 10 years in the two groups utilizing the EQ-5D quality of life questionnaire.
Angina Relief | 10 year follow-up
  Secondary aims include assessing angina status at 10 years in the two groups utilizing the Seattle Angina Questionnaire.

OTHER OUTCOMES:
Major adverse cardiac events | 10 year follow-up
  Additionally, we will compare individual rates of secondary clinical outcomes including myocardial infarction (MI), stroke, and repeat revascularization and combinations of the above, including death and MI, and death, MI, or stroke at 10-year follow-up after PCI or CABG.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fearon WF, Zimmermann FM, Ding VY, Takahashi K, Piroth Z, van Straten AHM, Szekely L, Davidavicius G, Kalinauskas G, Mansour S, Kharbanda R, Ostlund-Papadogeorgos N, Aminian A, Oldroyd KG, Al-Attar N, Jagic N, Dambrink JE, Kala P, Angeras O, MacCarthy P, Wendler O, Casselman F, Witt N, Mavromatis K, Miner SES, Sarma J, Engstrom T, Christiansen EH, Tonino PAL, Reardon MJ, Otsuki H, Kobayashi Y, Hlatky MA, Mahaffey KW, Desai M, Woo YJ, Yeung AC, Pijls NHJ, De Bruyne B. Outcomes after fractional flow reserve-guided percutaneous coronary intervention versus coronary artery bypass grafting (FAME 3): 5-year follow-up of a multicentre, open-label, randomised trial. Lancet. 2025 Apr 26;405(10488):1481-1490. doi: 10.1016/S0140-6736(25)00505-7. Epub 2025 Mar 30. PMID 40174598
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40174598/